CLINICAL TRIAL: NCT07380243
Title: Health Care by Food Planning Grant
Brief Title: Pathways to Prevention Food-is-Medicine Trial
Acronym: P2P
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Amrik Singh Khalsa (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); American Heart Association (Other); Ohio State University (Other)
Responsible Party: Sponsor-Investigator, Amrik Singh Khalsa, Principal Investigator, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: STUDY00005388; K23HL159312-04 (NIH)
Record Dates: First submitted 2025-12-19; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Heart Disease; Cardiovascular Health Status
Keywords: heart disease; cardiovascular
MeSH Terms: conditions — Heart Diseases | interventions — Nutrition Assessment

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Research coordinators who will be taking measurements from participants will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Nutrition Education only (Active Comparator): These participants will receive nutrition education only. All participants will receive nutrition education in this study, and other arms will be compared to this arm to assess the possibility that other conditions are more effective for improving cardiovascular health than education alone.
  Interventions: Behavioral: Nutrition Education
- Nutrition Education and Medically Tailored Groceries/Cooking Classes (Experimental): This group will receive nutrition education, medically tailored groceries, and cooking classes.
  Interventions: Behavioral: Nutrition Education; Behavioral: Medically tailored groceries/cooking classes
- Nutrition Education and PRO-CVH (Experimental): This arm will receive nutrition education and access to PRO-CVH, a web-based application designed to assess and communicate cardiovascular health.
  Interventions: Behavioral: Nutrition Education; Behavioral: PRO-CVH
- Nutrition Education and Healthy Conversational Skills (Experimental): This group will receive nutrition education and Healthy Conversational Skills, a brief behavior change counseling approach. Core principles include the clinician asking open-ended "What" and "How" questions, reflective listening, engaging in conversations that promote change, supporting the patient's autonomy in the change process, and goal-setting skills if the patient is ready
  Interventions: Behavioral: Nutrition Education; Behavioral: Healthy Conversation Skills
- Nutrition Education, Healthy Conversational Skills, and Medically Tailored Groceries/Cooking Classes (Experimental): Participants will receive nutrition education, Healthy Conversational Skills, medically tailored groceries, and cooking classes.
  Interventions: Behavioral: Nutrition Education; Behavioral: Healthy Conversation Skills; Behavioral: Medically tailored groceries/cooking classes
- Nutrition education, PRO-CVH, and medically tailored groceries/cooking classes (Experimental): This arm will receive nutrition education, access to PRO-CVH, medically tailored groceries, and cooking classes.
  Interventions: Behavioral: Nutrition Education; Behavioral: PRO-CVH; Behavioral: Medically tailored groceries/cooking classes
- Nutrition education, PRO-CVH, and Healthy Conversational Skills. (Experimental): Participants will receive nutrition education, access to PRO-CVH, and Healthy Conversational Skills.
  Interventions: Behavioral: Nutrition Education; Behavioral: PRO-CVH; Behavioral: Healthy Conversation Skills
- All Interventions (Experimental): Participants will receive nutrition education, access to PRO-CVH, Healthy Conversational Skills, medically tailored groceries, and cooking classes.
  Interventions: Behavioral: Nutrition Education; Behavioral: PRO-CVH; Behavioral: Healthy Conversation Skills; Behavioral: Medically tailored groceries/cooking classes

INTERVENTIONS:
Behavioral: Nutrition Education — Participants will receive handouts and access to an online curriculum for nutrition education. This education will be based on the Great Garden Detective Adventure (GDA) Team Nutrition, a USDA-supported Team Nutrition program that supports the United States Department of Agriculture (USDA) MyPlate guidelines and United States Dietary Guidelines. Educational content includes: increasing fruits and vegetables, improving whole grain intake, increasing water intake and limiting sugar-sweetened and high-fat beverages, selecting lean proteins, limiting sweets, and incorporating 60 minutes of physical activity per day.
Behavioral: PRO-CVH — PRO-CVH is the name of a cardiovascular health assessment and risk communication using a personalized, visual, and health-literacy friendly method. This web-based application is interactive and will assess and communicate cardiovascular health based on participant responses to surveys. The surveys will assess participant cardiovascular health indices based on the American Heart Association's Life's Essential 8 framework, behavioral components to change (e.g., motivation) and environmental barriers.
  Arms: All Interventions; Nutrition Education and PRO-CVH; Nutrition education, PRO-CVH, and Healthy Conversational Skills.; Nutrition education, PRO-CVH, and medically tailored groceries/cooking classes
Behavioral: Healthy Conversation Skills — Healthy Conversation Skills are a behavioral intervention where health coaches and participants engage in conversations that promote change, supporting the client's autonomy in the change process, and goal-setting skills
  Arms: All Interventions; Nutrition Education and Healthy Conversational Skills; Nutrition Education, Healthy Conversational Skills, and Medically Tailored Groceries/Cooking Classes; Nutrition education, PRO-CVH, and Healthy Conversational Skills.
Behavioral: Medically tailored groceries/cooking classes — Participants will receive funds for an online shopping cart, which will be tailored to promote a Mediterranean diet for cardiovascular health. Participants will attend cooking classes that use these foods. Classes are a skills-based training in home-cooked meals to educate parents on creating healthy meals on a budget. The curriculum consists of weekly classes by a Land Grant Extension Specialist. Each class includes nutrition education, hands-on cooking experience, and health promoting activities.
  Arms: All Interventions; Nutrition Education and Medically Tailored Groceries/Cooking Classes; Nutrition Education, Healthy Conversational Skills, and Medically Tailored Groceries/Cooking Classes; Nutrition education, PRO-CVH, and medically tailored groceries/cooking classes

SUMMARY:
The goal of this study is to learn whether combining healthy food access with personalized tools can help families improve heart health and make lasting lifestyle changes. The main questions the study aims to answer are:

* Do the new tools (PRO-CVH and Triple-C) help families improve their heart health?
* Which combination of tools and supports works best for families with limited access to healthy food?
* Is this type of program easy to carry out and acceptable to families and healthcare teams?

Families in the study will include one parent with a BMI greater than 30 who has Medicaid insurance and their child aged 6 to 11 years.

Depending on which group they are assigned to, families may:

* Receive food and nutrition education via handouts and/or online curriculum
* Have access to an online health assessment tool than can help you understand your/your child's risk factors for heart disease
* Work with a personalized health coach who can help you set goals for healthier living online/virtually.
* Receive medically tailored groceries and cooking classes.

Researchers will follow participants for several months to see how their heart health changes and which parts of the program work best together. The information from this study will help design a larger clinical trial to test a practical, cost-effective program that can help families build healthier habits and reduce their risk of heart disease.

DETAILED DESCRIPTION:
Heart disease is one of the leading causes of death in the United States and affects people from low-income communities at higher rates. Families with Medicaid insurance often face food insecurity, limited access to healthy foods, and other barriers that make it difficult to maintain a heart-healthy lifestyle. This study aims to address these challenges by combining nutrition support with behavioral tools that help families make and sustain healthy changes.

This study will test several "Food is Medicine" strategies that include medically tailored groceries, nutrition education, and new digital and communication tools to support healthier habits. The goal is to determine which combination of these strategies best improves heart health in parents and children.

The study will enroll families with one parent who has a body mass index (BMI) greater than 30, is enrolled in Medicaid, and has a child between 6 and 11 years old. The study focuses on this group because parents play a major role in shaping children's eating and activity habits. Supporting parents in making heart-healthy changes can improve the health of the whole family.

Participants will be assigned to different combinations of program components to see which are most effective and feasible. All families will receive some form of food and nutrition support, but each group may experience different combinations of the following components:

Food and Nutrition Education: Participants may receive educational materials or participate in an online course that covers healthy eating, cooking, and meal planning.

Online Health Assessment Tool (PRO-CVH): Families may have access to a digital tool that provides personalized feedback about heart health, based on the American Heart Association's Life's Essential 8 framework. This tool helps parents understand their current health status and identify areas for improvement.

Health Coaching: Some families will meet with a trained health coach or dietitian who can help set realistic goals, provide motivational support, and address barriers to change. Coaching will occur online or virtually.

Medically Tailored Groceries and Cooking Classes: Families may receive deliveries of heart-healthy groceries designed to support better cardiovascular health, along with cooking demonstrations to build practical food preparation skills.

The study will use a multiphase optimization design, which allows researchers to test multiple components together and identify the most effective and efficient combination. Because this is a pilot study, families will be followed for several weeks, with data collected at baseline and end of the study (4-8 weeks after enrollment).

Researchers will assess several outcomes, including:

* Changes in cardiovascular health indicators (such as blood pressure)
* Improvements in dietary patterns and readiness to change health behaviors
* Engagement with digital tools and counseling sessions
* Feasibility and acceptability of the intervention for families and healthcare teams

The information learned from this study will be used to plan a larger clinical trial. The ultimate goal is to design a scalable, cost-effective program that health systems and community organizations can use to help families build lasting heart-healthy habits.

By combining access to nutritious food with personalized tools and behavioral support, this research supports the American Heart Association's Health Care by Food initiative and its mission to reduce cardiovascular disease risk and promote longer, healthier lives.

ELIGIBILITY:
Inclusion Criteria:

* Parent or legal guardian of school-aged child (ages 6 - 11 years of age)
* Parent/legal guardian is 18 years or older and the primary caregiver at home
* Parent and/or child has an eligible Medicaid insurance plan
* Parent is able to read and speak English fluently
* Parent has BMI greater than 30 kg/m/m
* Ability to consume fruits and vegetables without concerns of any medication-nutrient interactions (for example, warfarin)

Exclusion Criteria:

* Parent not a legal guardian or the primary caregiver
* Non-English speakers
* Parent or child is diagnosed with active metabolic or digestive illnesses that may result in nutrient malabsorption (Crohn's disease, Celiac, irritable bowel syndrome, food allergies, etc.).

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular Health Behavior | pre-intervention and up to 8 weeks post-baseline
  A questionnaire will use participant responses to short-answer questions regarding lifestyle and dietary behaviors, physical activity, sleep, biological metrics, and nicotine exposure. The responses to this standardized questionnaire will result in a single composite score.
Intention to Change and Motivation to Change Lifestyle Behaviors | pre-intervention and up to 8 weeks post-baseline
  Self-reported survey to assess parent's intention to change their own and their child's lifestyle behaviors that put them at risk for future CVD.
Program Evaluation | up to 8 weeks post-baseline
  Survey to evaluate participant satisfaction with the intervention. The survey uses a 5-point Likert scale. There will be a series of statements and participants will select one of 5 responses ranging from 1 (completely disagree) to 5 (completely agree).
Qualitative Interviews | up to 8 weeks post-baseline
  Interviews with participants to assess participant thoughts on the intervention. Interviews will be analyzed qualitatively to learn about their experience with the intervention. Focus will be given to participant satisfaction.

SECONDARY OUTCOMES:
Perceived Benefits/Barriers of Change | pre-intervention and up to 8 weeks post-baseline
  Self-reported surveys to determine the perceived benefits and the perceived barriers to lifestyle change for themselves and their child.
Heart Disease Knowledge | Pre-Intervention
  Self-reported survey to determine an individual's knowledge of heart disease for themselves.
Adapted Risk Behavior Diagnosis (ARBD) Scale | pre-intervention and up to 8 weeks post-baseline
  A self-reported survey to assess perceived severity, perceived susceptibility, fear, anxiety, self-efficacy, and response efficacy with relation to parent and their perception of their child's future cardiovascular disease risk.
Self-reported Cardiovascular Disease Risk Factors | Pre-Intervention
  Surveys to determine parent's and their child's CVD risk factors.
Health Literacy | Pre-Intervention
  Measures to assess participant ability to understand health information. Questionnaire is a series of 5 questions about a nutritional label. Each participant response will be graded as "correct" or "incorrect" and will receive a score from 0 (no correct answers) to 5 (five correct answers).
Healthy Conversation Skills | Up to 8 weeks post-baseline
  All Healthy Conversation Skills will be recorded. All recorded calls will be compiled and used for data collection purposes. These recordings will be used to describe participant responses to Healthy Conversation Skills communication.
Childhood Opportunity Index | Pre-Intervention
  A measure that will map the quality of resources and conditions that matter for children to develop in a healthy way in the neighborhoods where they live.
Social Determinants of Health | pre-intervention and up to 8 weeks post-baseline
  Measures of social factors that may affect an individual's health and/or ability to change their lifestyle behaviors.
Attendance and Compliance | pre-intervention and up to 8 weeks post-baseline
  Attendance at all educational classes and scheduled encounters will be tracked.
Healthcare Use | pre-intervention and up to 8 weeks post-baseline
  Participants will be asked a series of questions about how many times they have accessed health care facilities. Participants will respond with a number. A higher number indicates a higher healthcare use.
Food Insecurity | pre-intervention and up to 8 weeks post-baseline
  Survey that asks participants a series of questions related to receiving assistance for food and difficulty accessing food. Questions about are asked as yes/no or as a 3-point Likert Scale ranging from 1 (often true) to 3 (never true).
Dietary Screener Questionnaire (DSQ) | pre-intervention and up to 8 weeks post-baseline
  Dietary Screener Questionnaire (DSQ) is a brief 26-item, semi-structured food frequency questionnaire.
Demographics | Pre-Intervention
  To help describe participant population, parent age, sex, race/ethnicity, level of education attainment, number of members in the household, and annual income will be recorded.
Participant Weight | pre-intervention and up to 8 weeks post-baseline
  Participants will be weighed, wearing light clothing and without shoes, on a standardized and calibrated digital scale. Weight will be recorded with a precision of 0.1 kg.
Bioelectrical Impedance | pre-intervention and up to 8 weeks post-baseline
  Calculation of body composition via bioelectrical impedance (e.g., InBody) which estimates free fat mass, muscle mass, fat mass and other body composition values.
Height | pre-intervention and up to 8 weeks post-baseline
  Participant standing height will be measured using a standardized fixed stadiometer with a vertical backboard and moveable headboard. Care will be taken to ensure that subjects are standing with feet and chin in proper position for the height measurement. Height will be recorded to the nearest 1 mm with shoes removed.
Body Mass Index (BMI) Percentile | pre-intervention and up to 8 weeks post-baseline
  BMI values are correlated with body fatness and are calculated using weight in kilograms divided by the square of height in meters. Based on the sex of the child, the correct BMI growth chart will be used. For children, the BMI percentile line closest to that point of intersection is the child's sex- and age-specific BMI percentile. For adults, BMI will be classified based on CDC criteria for normal weight, overweight, and obese.
Waist Circumference | pre-intervention and up to 8 weeks post-baseline
  Waist measurements will be completed for all participants using a tape measure. Waist circumference will be measured at the uppermost lateral border of the hip crest (ilium). Waist circumference will be measured with a precision of 0.1 cm per CDC guidelines for children and adults.
Blood Pressure | pre-intervention and up to 8 weeks post-baseline
  BP will be assessed by standard clinical methods using an Omron autocuff for all child and parent participants. Measurements will all be taken on the right side of the body unless the participant has a cast, amputation, or for some other reason the measurement cannot be taken on the right side.
Blood cholesterol | pre-intervention and up to 8 weeks post-baseline
  Cholesterol will be calculated via point-of-care methods using the Abbott Cholestex LDX machine. Standardized protocols as per Abbott will be used to collect the sample (using a 21-gauge pinprick needle and capillary tube) to collect the sample. The LDX machine will calculate the cholesterol within 5-10 min.
Blood glucose | pre-intervention and up to 8 weeks post-baseline
  3-month average glucose will be estimated via hemoglobin A1c using the Abbott Affinion machine. Standardized protocols as per Abbott will be used to collect the sample (using a 21-gauge pinprick needle and capillary tube) to collect the sample. The Affinion machine will calculate the hemoglobin A1c within a few minutes.

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided